Title: Repeated TMS at Low Frequencies to Reduce Seizure

NCT Number: NCT03154307

Protocol Number: 15-135

Document Date: September 21, 2021

#### I. SUMMARY OF THE RESEARCH

Perform non-invasive neuro-navigated repeated Transcranial Magnetic Stimulation (rTMS) at low frequencies (LF) with the intent to reduce the occurrence of seizures over time. Seizure reduction and improvements in the quality of life in patients with epilepsy will be associated with increased cortical inhibition resulting from the LF-rTMS sessions over time. This procedure using rTMS at low frequencies (LF-rTMS) between 0.5 and 1 Hz is a safe and painless method for noninvasive focal cortical brain stimulation, which will be evaluated in its efficacy at reducing/suppressing seizures. Accordingly, we propose a clinical trial in patients with epilepsy to test whether LF-rTMS can improve seizure suppression. The location of the presumed 3D source in the brain will be stimulated for few minutes (10 to 15mns). With the same rTMS modality, we will also perform motor threshold mapping in conjunction with its fully integrated and compatible electroencephalography (EEG) module.

Despite the progress made in the development of multimodal imaging algorithms, there are still limitations and drawbacks to be overcome in the area of time and space alignments. The simultaneous use (time alignment) of different recording modalities on a same patient (space alignment) would validate a given outcome as long as it is imaged or recorded in more than one imaging/recording modality. As such, brain mapping and 3D source localization are consolidated in a same 3D space and in context to the 3D source where seizures are anticipated to emanate from. The multimodality structure relies in the simultaneous use of TMS, MRI, EEG and Electromyography (EMG), all non-invasive, safe, and FDA approved. The complete procedure will include tasks of motor threshold mapping using non-invasive brain navigated magnetic stimulation, while simultaneously monitoring EEG and EMG. The study is of minimal risk with common risks/discomforts of the test limited to mild and brief discomfort of the skin on the scalp from the Velcro strap or the EEG electrodes. Also, occasional side effects of the test are minor and brief headache from prolonged TMS stimulation.

The significance of this work is related to addressing the effectiveness of long-term use of rTMS for medically refractory patients (failed two or more medications) as a non-invasive alternative to other established techniques (i.e. VNS, RNS, among others). For this purpose, we will unify data from different sources whose analysis and results are strengthened and validated in more than one modality (TMS, MRI, EEG in consortium), which will secondarily provide higher resolution for assessing the dysfunction in both temporal and spatial domains. All of these steps are to ensure the delivery of the most effective rTMS brain stimulation with the intent to reduce/suppress the occurrence of seizures in patients with epilepsy to include both children and adult populations.

### II. SCIENTIFIC BACKGROUND & LITERATURE REVIEW

Transcranial Magnetic Stimulation with both single (sTMS) and repetitive simulation (rTMS) capabilities is a non-invasive technology, which serves not only as a powerful tool for mapping the eloquent cortex of the brain, but provides great potential for treatment and eliciting new insights into a variety of brain disorders, especially for patients who do not benefit from drug treatments. The TMS technology was introduced in the 1980s, and since then, it has been used in clinical care for several neurological disorders [1–4]. The initial intent of this technology was to improve the health of patients with depression as exemplified in studies [5–8]. Its application has now been

extended to gauge the merits of magnetic stimulation to other neurological disorders such as epilepsy [9–11], Huntington's disease [12], Parkinson's disease [13], different effects of schizophrenia [14–16], Alzheimer's disease, and effects of aging [17, 18], in patients who have had a stroke [19–21], autism [22, 23], and attention deficit and hyperactivity disorders [23, 24]. These are by no means an exhaustive listing of such noteworthy references, but these are examples of studies that highlight the extensive use of TMS technology. It should be noted that the use of TMS can be performed under two modes of operation, namely, single pulse [25] or repetitive mode of stimulation [26, 27].

The hypothesis is that low frequency brain stimulation focused on and around the seizure onset zone will reduce the occurrence of seizures over time. We base this hypothesis on clinical trials and reports on the treatment of seizures reported in the literature. It has been shown that high frequency rTMS, although beneficial in the treatment of patients with depression, can actually cause seizures [28], while low-frequency rTMS has the opposite effect in that it can actually inhibit the occurrence of such seizures. Modulating brain activity is shown to depend on the selection of the frequency used during stimulation [29, 30]. Therefore, and on the basis of this knowledge, we will restrict the brain stimulation process to a low frequency range between 0.5 and 1 Hz rTMS in people with focal and generalized epilepsy, while taking into consideration all the safety guidelines, ethical issues, and required precautions from prior research in the use of TMS technology [31, 32, 33].

The significance of this work is to address the efficacy of the long-term use of rTMS in the treatment of refractory epilepsy patients. Additionally, the integration of multimodal imaging where TMS, MRI, and EEG could provide data not available through DCS or fMRI alone, which in turn can only augment our understanding of brain mapping and brain dynamics. This study will employ a carefully planned low frequency rTMS protocol, with therapeutic sessions over a one-year time frame, with a possible extension phase protocol if initial study is successful.

### **III.RESEARCH OBJECTIVES**

- 1. To reduce/suppress the number of seizures in patients with medically intractable epilepsy (partial and generalized) with the use of long-term LF-rTMS. Stimulation will be applied with determined seizure onset zone by inverse solutions and 3D software algorithms of analysis of electroencephalographic data. This objective is based on promising rTMS studies that reported reductions in seizure frequency. The primary continuous outcome measures for this aim will be seizure frequency, EEG epileptiform discharge frequency, seizure severity scale, and psychometric testing.
- 2. Statistical analysis will be conducted using ANOVA and secondary outcome measures will analyze the number of patients whose seizure frequency decreases by at least 50% (e.g., the "responder" threshold used in studies of anticonvulsant efficacy).
- 3. Localize through TMS stimulation motor threshold cortex mapping of the abductor pollicus brevis-evoked response. This is an important step for determining the appropriate patient-specific stimulation threshold.
- 4. Measure EEG alpha asymmetry before and after rTMS and compare the change in this continuous variable among treatment and sham groups in intractable epilepsy. We

hypothesize, that rTMS will alter the ratio of right to left EEG alpha power (8-13 Hz). Alpha asymmetry is known to be common in patients with epilepsy in contrast to healthy controls where alpha symmetry is seen as more prevalent.

#### IV. INCLUSION AND EXCLUSION CRITERIA

All individuals between ages 18 to 80 that are medically refractory who have completed informed consent/assent, and able to cooperate with non-sedated navigated TMS testing will be included. Exclusion criteria include the presence of implanted electronic devices (e.g., pacemaker, medication pump, brain or vagus nerve stimulator, cochlear implant), intracranial metal (e.g., aneurysm clip), or inability to cooperate with the rTMS session.

Goal recruitment will be 90 epilepsy patients, based on the following:

- At least 3 seizures in one month
- No status epilepticus for 1 year
- No change in medication for 1 month

#### V. METHODS AND ACTIVITIES

#### 5.1 Interventions and Interactions of the Research Study

An Informed Consent will be obtained by Baptist Health personnel and the subject will be explained the aims and procedures of the research task that will be performed by FIU personnel.

- Positioning of the subject in the TMS chair along with the registration apparatus (spectacles or head band) and performing a high-resolution (< 2mm) registration of the subject head to the pre-acquired magnetic resonance imaging (MRI) since the TMS machine is MRI-guided.
- Connecting 1-6 EMG surface electrodes on target muscles to evaluate muscle response to TMS stimulation, and
- EEG electrodes will be placed according to the 10-20 system montage.

The systems (EMG and EEG) will continuously record the activity from the subject throughout the procedure. It should be noted that since these acquisition techniques, which are completely non-invasive and used regularly in clinical settings, render little or no discomfort to the test subjects. There will be a neurologist (Dr. Alberto Pinzon) on the premises during all procedures. Sections 5.1-5.3 and 5.4.3-5.4.4 of the "Methods and Activities", as explained below will be performed completely by FIU personnel (Mercedes Cabrerizo, Ph.D. and Ms. Niovi Rojas). Malek Adjouadi, Ph.D. from FIU will supervise all the protocol outcomes. Dr. Pinzon will refer all epileptic patients that will be included in this study research. Also copies of standard care MRI images (not taken as part of this study) will be provided by Baptist Hospital Radiology Department after enrolled subjects sign a HIPAA agreement to allow it.

### 5.2 TMS mapping and recording

The technology used in this research study is based on the so-called Neuro-navigated Brain Stimulation (NBS), a technology developed for mapping the eloquent cortex of the brain as well for therapy as currently used on different neurological disorders in different centers and healthcare

providers. This newly acquired technology by the CATE center is to improve accuracy in the diagnosis and in improving mapping the brain non-invasively. TMS mapping and recording will allow for (1) MRI-guided neuro-navigation with electric-field controlled stimulation to precise 3D targets in the cortex; (2) powerful and highly focal magnetic stimulator and coils with the ability to monitor the point of focality as well depth attenuation; (3) a compatible fully integrated EMG for motor functions; and (4) a compatible 60-channel EEG module for integrating brain electrical activities at rest and under the TMS stimulation process. TMS thus offers a non-invasive alternative to DCS (gold standard). This can be further augmented with the fMRI images in order to validate the location of these eloquent cortical areas.

Since the TMS is FDA approved for motor threshold mapping, the following protocol is used to map the eloquent cortex.

### 5.2.1 Motor Threshold Mapping Protocol

All the patients will lie down in a comfortable chair in a supine position. The Nexstim system's 6-channel EMG module (SR=1450 Hz, cut-off frequency of 350 Hz for the low pass filter) will automatically calculate the motor evoked potential (MEP) amplitudes and latencies as the motor cortex (cortex area of the thumb) is stimulated. Disposables Ag-AgCL surface electrodes will be used to record the MEP responses displayed in a computer screen in order to assess the validity of the response based on the strength of MEPs, reflecting the ability of that area to develop a muscle contraction.

This protocol will consist of the following two steps:

- Perform TMS in order to determine the motor threshold for each individual patient.
- In order to obtain the motor threshold, the intensity of the TMS is gradually increased in order to elicit responses from the Abductor Pollicis Brevis (APB) muscle near the thumb.
- Once the motor threshold is determined the complete tracking of the motor cortex is carried out at an intensity of 10% greater than the motor threshold.
- The entire process of motor cortex mapping is estimated to take 15-20 minutes.

Prior studies have demonstrated that partial motor threshold can vary in a person from session to session and for this reason, it will be performed every time patients are treated.

### 5.3 Epilepsy Protocol for rTMS at low frequencies in Epilepsy (long-term protocol)

Repetitive transcranial magnetic stimulation (rTMS) at low frequency range (0.5-1 Hz), LF-rTMS is a safe and painless method for noninvasive focal cortical brain stimulation which is efficacious in suppressing seizures. Accordingly, we propose a clinical trial in patients with epilepsy to test whether LF-rTMS can improve seizure reduction/suppression. The location of the presumed 3D source in the brain and its immediate surroundings will be stimulated for 14 minutes at these low frequencies.

Existing protocols that are related to this work [34-41] are listed in Table 1. These were reviewed in order to bring in synergy the strengths of each for carrying out safe and effective rTMS sessions. Accordingly, we propose a long term trial in patients with focal and generalized epilepsy, to test whether LF-rTMS can reduce/suppress the occurrence of seizures, and determine for how long such outcomes can last for each patient. The proposed protocol that will be followed in this study is described in Table II on the basis of the knowledge gained from these previous studies.

**Table 1**: Existing Protocols.

| Cited<br>Literature | Frequency | Threshold | Stimuli | Schedule | Coil | Outcome-<br>seizures | Position | Daily<br>Stimulation<br>time |
|---|---|---|---|---|---|---|---|---|
| Cantello,<br>et al.<br>2007 [34] | 0.3 Hz | 100%MT<br>65%MSO | 500/trai<br>n | trains/day For 5 days | 0 | No change | vertex | 28 min. |
| Fregni, et al. 2006 [35] | 1Hz | 70%MSO | 1200/tra<br>in | 1<br>train/day<br>For 5<br>days | 8 | Decreasing | 3D<br>source<br>vertex | 20 min. |
| Theodore<br>, et al.<br>2002 [36] | 1 Hz | 120% MT | 900/trai<br>n | trains/day For 1 week | 8 | Decreasing | 3D<br>source | 15 min. |
| Tergau,<br>et al.<br>2003 [37] | 0.33, 1 Hz | Below MT | 1000/Tr<br>ain | 1<br>train/day<br>For 5<br>days | 0 | Decreased<br>0.33 Hz | vertex | 55 min.<br>17 min. |
| Brasil-<br>Neto, et<br>al. 2004<br>[38] | 0.5 Hz | 90% MT | 100/trai<br>n | Biweekly<br>/ 4 weeks | 8 | Decreased | 3D<br>source<br>vertex | 3 min. |
| Misawa,<br>et al.<br>2005 [39] | 0.5 Hz | 90%MT | 100 | Single<br>session<br>repeated<br>at 3<br>months | 8 | Decreased<br>for 2<br>months | 3D<br>source | 3 min. |
| Menkes,<br>et al.<br>2000 [40] | 0.5 Hz | 95%MT | 20/train | 5<br>trains/day<br>Biweekly<br>for 3<br>months | 0 | decreased | 3D source | 0.6 min. |
| Rossi, et<br>al. 2004<br>[41] | 1 Hz | 90% rMT | 900 | Single session | 8 | decreased | 3D<br>source | 15 min. |

MT: Motor threshold, MSO: Maximum stimulator output

**Table 2**: Suggested Long-Term Protocol for this Study: Treatment vs. Placebo Groups (Stimulation time: 14 minutes)

| Frequency | Threshold | Stimuli | Schedule | Coil | Position | Study |
|-----------|-----------|---------|----------|------|----------|-------|

| | | | | | | Design |
|---|---|---|---|---|---|---|
| 1Hz | 120%MT | 800 | 5 days/week for 2<br>weeks<br>1/week for 1 month<br>1/month for 11<br>months | 8 | 3D Source<br>Localization,<br>vertex, and bipolar<br>frontal | double-<br>blinded, sham-<br>controlled |
| 1Hz | 120%MT | 800 | 5 days/week for 2<br>weeks<br>1/week for 1 month<br>1/month for 11<br>months | 8 | coil will be placed<br>with an angle of 45<br>degrees with<br>respect to the<br>scalp without<br>direct contact | double-<br>blinded, sham-<br>controlled |

Using a single-blinded, sham-controlled design, we will screen patient's age 2 to 80 years with focal and generalized retractable epilepsy. Baseline data will include a detailed seizure diary over 4 weeks, psychometric testing/neuropsychology evaluation, and 20-minute EEG recordings. Each patient will then begin treatment with 14 minute sessions of 1 Hz rTMS or sham rTMS, 120%MT, and 800 stimuli on the position of the calculated 3D source using EEG, MRI, and digitized electrode locations. The protocol will be divided in 3 groups (Groups 1, 2 and 3) as follows:

- Groups 1, 2, and 3: LF-rTMS for 2 weeks (5 days per week for total of 10 days).
- Group 1: protocol total duration: 1 year: LF-rTMS 1 session/week for 1 month (4 days), and LF-rTMS 1 session/month for 11 months
- Group 2: protocol total duration: 1 year: LF-rTMS 1session/month for 12 months
- <u>Group 3 (placebo protocol, total duration: 1 year)</u>: LF-rTMS 1session/week for 1 month (4 days); and LF-rTMS 1session/month.

During each session EEG will be recorded. Also, we would update number of events and frequency data from ongoing seizure diary. Psychometric testing will be performed at the beginning of study, 3 months, and at the end of the study. Thus, each patient will have rTMS testing, psychometrics, and EEG recordings.

Goal recruitment will be 90 medically refractory participants, with 30 participants for each of the three groups, based on the following:

- At least 3 seizures in one month
- No status epilepticus for 1 year
- No change in medication for 1 month

In retrospect, promising rTMS studies have reported reductions in seizure occurrence [35, 42-54]. Several studies [45-48] included children, and reported improvement in seizure occurrence in the majority of these children, due to a modulation in cortical excitability, induced by low frequency rTMS. Other studies measured EEG alpha asymmetry [49] before and after rTMS to assess the change in this continuous variable among treatment and sham groups in intractable epilepsy. In these studies, it is hypothesized that rTMS could alter the ratio of right to left EEG alpha power

(8-13 Hz). Alpha asymmetry is known to be present in patients with epilepsy in contrast to healthy controls. The major objective in all of these studies is to seek seizure reduction associated with increased cortical inhibition resulting from the LF-rTMS sessions [34, 50-53]. TMS (single or repetitive pulse) thus offers a noninvasive option that could serve as a therapeutic tool that will reduce the occurrence of seizures.

## 5.3.1 Epilepsy Protocol for rTMS at low frequencies in Epilepsy (short-term protocol)

Epilepsia partialis continua (EPC) can be considered the status epilepticus (SE) equivalent of focal onset seizure with retention of awareness. EPC may occur as a single episode, repetitive episodes, and it may be chronic progressive or non-progressive. The significance of this work is to address the efficacy of the short-term use of rTMS in the treatment of EPC patients. This study will employ a carefully planned low frequency rTMS protocol, with therapeutic sessions over a short period of time (3 to 5 days), with a possible extension phase protocol if initial study is successful.

Existing protocols that are related to this work [1-7] are listed in Table 3. These were reviewed in order to bring in synergy the strengths of each for carrying out safe and effective rTMS sessions. Accordingly, we propose a short term trial in patients with EPC, to test whether LF-rTMS can reduce/suppress the status epilepticus, and determine for how long such outcomes can last for each patient. The proposed protocol that will be followed in this study is described in Table 4 on the basis of the knowledge gained from these previous studies.

During each session EEG will be recorded. Goal recruitment will be 10 acute phase medically refractory participants, based on the following:

- At least 2 medications failed
- At least 24 hours of acute phase
- Family consent or available proxy (legal representative)

### Equipment:

The MagVita TMS is CE approved for "treatment of Major Depressive Disorder. MagVenture's rTMS system is effective and it is an alternative to medications.

| Cited<br>Literature | Frequen<br>cy | Threshold | Stimuli | Schedule | Coil | Outcome-<br>seizures | Position | Stimulation time |
|---|---|---|---|---|---|---|---|---|
| Gersner, et al. 2016 (1) | 20Hz | 80%MO | 500/train | 10 trains<br>of 3s with<br>30s<br>intertrain<br>One time | 8 | Reduced epileptic spike frequency decreased seizures during stimulation | vertex | Single<br>5 min. |

**Table 3**: Existing Protocols.

| Liu A, et al.<br>2015 (3) | 1Hz | 70%MO | | 1 train | 8 | Reduced<br>epileptic<br>spike<br>frequency<br>and seizures | 3D source | 20 min. |
|---|---|---|---|---|---|---|---|---|
| Rotenberg,<br>2009 (4) | 1Hz:1800<br>sec. | 100%MT | 3 trains | 3 trains | | Seizures<br>stopped | 3D<br>source | 1800 sec |
| Graff Guerrero. 2004(5) | 20Hz | 50%MO | 15 trains | 15 trains of 2 sec | | Seizures<br>stopped | 3D source | |
| Graff Guerrero. 2004(5) | 20Hz | 128%MT | 15 trains | 15 trains of 2 sec | | Improved<br>EEG | 3D source | |
| Schrader<br>LMKL,<br>2005 (6) | 0.5 Hz | 100%MT | 16 trains<br>of 900<br>sec | 2 trains<br>per<br>session,<br>biweekly,<br>for 4<br>weeks) | | decreased<br>seizures | 3D source | |
| Misawa S,<br>2005 , (7) | 0.5 Hz | 90%MT | 1 train<br>of 200<br>sec | 1 train | | Seizures<br>stopped | 3D source | |

MT: Motor threshold, MSO: Maximum stimulator output

 Table 4: Suggested short-Term Protocol for this Study: (Stimulation time: minutes)

| Frequency | Threshold | Stimuli | Schedule | Coil | Position | Study<br>Design |
|---|---|---|---|---|---|---|
| 1Hz | 100%MO | | Up to 5 days/ | 8 | 3D Source<br>Localization or<br>vertex | Open-label |

## **5.3.2** Limitations and Alternative Approaches

While TMS is a safe, painless, technically easy procedure, because the orientation of the magnetic field of stimulation needs to be perpendicular to the electrical field of stimulation, TMS may not always generate a response. In such a case, the benefit of the stimulation technique may be limited. The abductor pollicis brevis (APB) is a low voluntary recruitment threshold motor unit, easily activated in most individuals using TMS. However, should this fail to activate with maximal stimulation, another muscle of similar threshold can be substituted: either the first dorsal interosseous or the abductor digiti minimi. These muscles are all in the palm of the hand.

### 5.3.3 Emergency Response and Treatment Protocol in case of Seizure

A neurologist (Dr. Alberto Pinzon) will be on the premises at all times during the rTMS treatment. In the immediate vicinity of the TMS machine where the patient is laying down on a comfortable chair similar to the ergonomic dental chair, no harmful objects will be present. In case a patient suffers the occurrence of a seizure during an rTMS session, the following steps are undertaken:

- Code rescue will be initiated for the management of acute seizure for patient safety according to hospital's protocols and as below.
- Diastat AcuDial (diazepam rectal gel) will be kept at the chair side in case any seizures are
  provoked. DIASTAT is a gel formulation of diazepam intended for rectal administration
  in the management of selected, refractory patients with epilepsy, on stable regimens of
  AEDs, who require intermittent use of diazepam to control bouts of increased seizure
  activity for patients 2 years and older.
- If a seizure occurs, testing (TMS) will be postponed at least 1 hour, or until baseline function returns.
- Patient will be placed on their left side in the recovery position to promote airway and prevent aspiration.
- Harmful objects will be moved out of the way, head will be protected.
- Patient will not be restrained. Objects will not be placed in the mouth. Adequate ventilation will be ensured.
- Respiratory changes such as skin color increase/decrease in respiratory rate and noisy or congested breathing will be monitored. If the patient is not breathing, rescue breathing will be started immediate medical attention will be followed. Suction apparatus, clean gloves and pillows will be available for immediate use.

http://www.epilepsy.com/get-help/staying-safe and http://www.epilepsy.com/get-help/managing-your-epilepsy.http://www.emergencycareforyou.org/EmergencyManual/WhatToDoInMedicalEmergency/Default.aspx?id=268.http://www.webmd.com/epilepsy/epilepsy-seizure-what-to-do-in-an-emergency

### **5.4 Multimodal Imaging**

This TMS based protocol for epilepsy relies on multimodal imaging to benefit from (1) structural MRI for MRI-guided TMS motor threshold mapping and for situating in context the 3D source of seizure onsets; and (2) EEG for determining the 3D source exploiting the presence, positioning and singular nature of the interictal spike waveforms.

### **5.4.1 Magnetic Resonance Imaging -MRI**

All patients that will undergo TMS brain stimulation would have had both magnetic resonance imaging (MRI) recording done at any of our collaborating hospitals (Miami Children's Hospital, Baptist Hospital or other) as it concerns this study. Since TMS is an MRI-guided machine, its use in conjunction with an MRI of a patient, it becomes possible to perform pinpointed navigated mapping of the language and motor areas of the brain. And when a 3D source is determined using interictal spikes of the EEG, such a source is also rendered in the context of the 3D brain of the patient.

### 5.4.3 Electroencephalography recordings - EEG

EEG recordings will be performed using the XLTEK EEG (Electroencephalograph) system. EEG signals will also be collected before and after some selected rTMS sessions, so that more comprehensive subject-specific connectivity maps could be obtained [54-57]. This is performed in order to assess the connectivity maps as a function of the determined position of the 3D source.

This system will be used to record the brain's spontaneous electrical activity and evoked responses non-invasively from the scalp. XLTEK EEG is a robust whole-head EEG system that can be used to record EEG activity so as to determine the 3D source of seizures on the basis of interictal spikes, or subsequent to this first step. Some of the research themes that will be investigated include (1) EEG activity analysis on the basis of the cortical and sub-cortical stimulation using repetitive pulse TMS (rTMS); (2) Study the functional connectivity between areas and the changes that occur in the brain before and after stimulating motor and language areas, respectively; (3) assess TMS-induced modulation of brain rhythms with respect to rest state.

Also EEG recordings in some cases may be performed using the Nexstim eXimia EEG system, designed specifically to be fully compatibility with the TMS machine, and is another major component that can be purchased alongside the TMS machine, which we did. *It is important to note that with the new TMS technology, an EEG module is fully integrated, and unlike the inherent noise in the integration of EEG and fMRI, both EEG and TMS signals are fully compatible as the TMS does not affect the EEG signal.* Consequently, EEG signals will also be collected during brain mapping, so that more comprehensive subject-specific connectivity maps could be obtained [54-57]. This is performed in order to assess the connectivity maps as a function of the determined position of the 3D source.

#### 5.5. Risks Associated with the Recording Modalities

#### **5.5.1 Risks of TMS**

TMS often causes minor short-term side effects. These side effects are generally mild and typically improve after the first week or two of treatment. They can include:

- Headache.
- Scalp discomfort at the site of stimulation.
- Tingling, spasms or twitching of facial muscles.
- Lightheadedness.
- Discomfort from noise during treatment
- Mild and brief discomfort of the skin on the scalp from the Velcro strap or the EEG electrodes.

#### Uncommon side effects include:

- Mild and brief headaches or neck aches from the TMS stimulation. Serious side effects are rare. They can include:
- Seizure occurring during TMS stimulation at high frequencies. This has only been known to happen in 1% of children and adults with epilepsy, and in less than 1% of children and adults without epilepsy.

- Mania, particularly in people with bipolar disorder.
- Hearing loss due to inadequate ear protection during treatment.

#### 5.5.3 Risks of EEG recording

There are no known risks for this standard noninvasive scalp EEG recordings, except for slight discomfort due to the placement of some of the electrodes that may be too tight on the scalp.

## 5.5. 3 Minimizing Risks, Harms, and/or Discomforts

In order to reduce discomfort due to use of EEG electrodes, 'comfort rings' are used. As for rTMS stimulation, a mechanical arm with several degrees of freedom is designed to hold the TMS coil to eliminate any potential for pressure on the head of the subject, something that could happen if the coil were handheld by the clinician.

Previous studies have demonstrated that motor threshold mapping in normal subjects is not associated with provoking seizures [58].

#### VI. DATA TO BE COLLECTED AND DATA ANALYSIS PROCEDURES

Patients will be given a questionnaire to fill out their demographic and health information. Original medical records may be requested and stored by primary neurologist.

For each patient, the following types of data will be collected:

- A 3D MRI volume: This high resolution volumetric imaging data will be collected so that the final results could be displayed in concordance with the regions that were found to be active according to the task applied (motor or speech).
- Scalp EEG s in order to extract time and frequency domain parameters to assess the reaction of the brain to magnetic stimulation using different intensities and frequencies. The lateralization index will be calculated to define the dominant cerebral hemisphere for the language task.
- DICOM stimulation maps for motor threshold mapping.
- EMG data obtained from 1-6 EMG electrodes used for monitoring different muscle groups.

The data will be collected and stored for each patient undergoing the study. All the data will be de-identified by converting into alphanumeric values. The encoded values will be stored in password-protected servers accessible only to research personnel (FIU/Baptist) with authorization throughout data collection and analysis.

All identifiers will be removed from the data once they are transferred off the TMS computer and gathered into a pooling database, where each case will have a unique consecutive identification number. This information will be annotated in a separated document kept in the office of the PI (Dr. Pinzon).

Statistical analysis will be conducted using SPSS 14.0 software. The baseline seizure frequency and seizure frequency change after treatment will be computed from average weekly seizure frequencies before and after rTMS treatment for each patient. A patient data will be categorized into two treatment groups: rTMS treated and placebo groups.

#### VII. DESCRIPTION OF WRITTEN CHILD/ADULT CONSENT PROCESS

At a potential subject's visit to the physician's office or hospital, the investigator(s) will provide a comprehensive explanation of the purpose, procedures, possible risks/benefits of the study, and participant responsibilities, and discuss the fact that his/her participation is voluntary, that he/she may withdraw from the study at any time, and that the decision not to participate or to withdraw will not affect his/her regular medical care. Potential participants or their surrogates will be given ample opportunity to ask questions and to consider their decision. If the subject or the surrogate agree to participate, then a signed and dated written informed consent will be obtained.

A copy of the consent form will be given to the participant or the surrogate, and another copy will be placed in the subject's medical record. The informed consent form will be obtained by the investigators listed to perform informed consent procedures.

#### VIII. EXTENSION PHASE

If the results from this study demonstrate significant medical improvement, patients will be offered an extension phase where they could continue receiving the same parameters of stimulation for one to two additional years at no expense

### **REFERENCES**

- [1] M. Kobayashi and A. Pascual-Leone, "Transcranial magnetic stimulation in neurology," *Lancet Neurology*, vol. 2, pp. 145-156, Mar 2003.
- [2] M. Hallett, "Transcranial magnetic stimulation and the human brain," *Nature*, vol. 406, pp. 147-150, Jul 13 2000.
- [3] P. M. Rossini and S. Rossi, "Transcranial magnetic stimulation: diagnostic, therapeutic, and research potential," *Neurology*, vol. 68, pp. 484-8, Feb 13 2007.
- [4] H. R. Siebner, G. Hartwigsen, T. Kassuba, and J. C. Rothwell, "How does transcranial magnetic stimulation modify neuronal activity in the brain? Implications for studies of cognition," *Cortex*, vol. 45, pp. 1035-1042, Oct 2009.

- [5] K. Udupa, T. N. Sathyaprabha, J. Thirthalli, K. R. Kishore, T. R. Raju, and B. N. Gangadhar, "Modulation of cardiac autonomic functions in patients with major depression treated with repetitive transcranial magnetic stimulation," *J Affect Disord*, vol. 104, pp. 231-6, Dec 2007.
- [6] Fox, Michael D.; Liu, Hesheng; Pascual-Leone, Alvaro, "Identification of reproducible individualized targets for treatment of depression with TMS based on intrinsic connectivity", NeuroImage, vol. 66, pp. 151-160, February 2013.
- [7] C. Plewnia, P. Pasqualetti, S. Grosse, S. Schlipf, B. Wasserka, B. Zwissler, and A. Fallgatter, "Treatment of major depression with bilateral theta burst stimulation: A randomized controlled pilot trial," *Journal of Affective Disorders*, vol. 156, pp. 219-223, Mar 2014.
- [8] E. V. Harel, A. Zangen, Y. Roth, I. Reti, Y. Braw, and Y. Levkovitz, "H-coil repetitive transcranial magnetic stimulation for the treatment of bipolar depression: an add-on, safety and feasibility study," *World Journal of Biological Psychiatry*, vol. 12, pp. 119-126, Mar 2011.
- [9] E. H. Bae, L. M. Schrader, K. Machii, M. Alonso-Alonso, J. J. Riviello, Jr., A. Pascual-Leone, and A. Rotenberg, "Safety and tolerability of repetitive transcranial magnetic stimulation in patients with epilepsy: a review of the literature," *Epilepsy & Behavior*, vol. 10, pp. 521-8, Jun 2007.
- [10] A. Ponnusamy, J. L. Marques, and M. Reuber, "Comparison of heart rate variability parameters during complex partial seizures and psychogenic nonepileptic seizures," *Epilepsia*, vol. 53, pp. 1314-21, Aug 2012.
- [11] P. R. Bauer, S. Kalitzin, M. Zijlmans, J. W. Sander, and G. H. Visser, "Cortical Excitability as a Potential Clinical Marker of Epilepsy: A Review of the Clinical Application of Transcranial Magnetic Stimulation," *International Journal of Neural Systems*, vol. 24, Mar 2014.
- [12] A. L. Philpott, P. B. Fitzgerald, T. D. R. Cummins, and N. Georgiou-Karistianis, "Transcranial magnetic stimulation as a tool for understanding neurophysiology in Huntington's disease: A review," *Neuroscience and Biobehavioral Reviews*, vol. 37, pp. 1420-1433, Sep 2013.
- [13] F. Fregni, C. M. Santos, M. L. Myczkowski, R. Rigolino, J. Gallucci-Neto, E. R. Barbosa, K. D. Valente, A. Pascual-Leone, and M. A. Marcolin, "Repetitive transcranial magnetic stimulation is as effective as fluoxetine in the treatment of depression in patients with Parkinson's disease," *Journal of Neurology Neurosurgery and Psychiatry*, vol. 75, pp. 1171-1174, Aug 2004.

- [14] R. Prikryl, L. Ustohal, H. P. Kucerova, T. Kasparek, J. Jarkovsky, V. Hublova, M. Vrzalova, and E. Ceskova, "Repetitive transcranial magnetic stimulation reduces cigarette consumption in schizophrenia patients," *Progress in Neuro-Psychopharmacology & Biological Psychiatry*, vol. 49, pp. 30-35, Mar 3 2014.
- [15] Y. Levkovitz, L. Rabany, E. V. Harel, and A. Zangen, "Deep transcranial magnetic stimulation add-on for treatment of negative symptoms and cognitive deficits of schizophrenia: a feasibility study," *Int J Neuropsychopharmacol*, vol. 14, pp. 991-6, Aug 2011.
- [16] M. Frantseva, J. Cui, F. Farzan, L. V. Chinta, J. L. P. Velazquez, and Z. J. Daskalakis, "Disrupted Cortical Conductivity in Schizophrenia: TMS-EEG Study," *Cerebral Cortex*, vol. 24, pp. 211-221, Jan 2014.
- [17] P. Julkunen, A. M. Jauhiainen, S. Western-Punnonen, E. Pirinen, H. Soininen, M. Kononen, A. Paakkonen, S. Maatta, and J. Karhu, "Navigated TMS combined with EEG in mild cognitive impairment and Alzheimer's disease: A pilot study," *Journal of Neuroscience Methods*, vol. 172, pp. 270-276, Jul 30 2008.
- [18] P. M. Rossini, S. Rossi, C. Babiloni, and J. Polich, "Clinical neurophysiology of aging brain: From normal aging to neurodegeneration," *Progress in Neurobiology*, vol. 83, pp. 375-400, Dec 2007.
- [19] F. C. Hummel and L. G. Cohen, "Non-invasive brain stimulation: a new strategy to improve neurorehabilitation after stroke?," *Lancet Neurology*, vol. 5, pp. 708-712, Aug 2006.
- [20] N. Yozbatiran, M. Alonso-Alonso, J. See, A. Demirtas-Tatlidede, D. Luu, R. R. Motiwala, A. Pascual-Leone, and S. C. Cramer, "Safety and behavioral effects of high-frequency repetitive transcranial magnetic stimulation in stroke," *Stroke*, vol. 40, pp. 309-12, Jan 2009.
- [21] F. Fregni, P. S. Boggio, A. C. Valle, R. R. Rocha, J. Duarte, M. J. Ferreira, T. Wagner, S. Fecteau, S. P. Rigonatti, M. Riberto, S. D. Freedman, and A. Pascual-Leone, "A sham-controlled trial of a 5-day course of repetitive transcranial magnetic stimulation of the unaffected hemisphere in stroke patients," *Stroke*, vol. 37, pp. 2115-22, Aug 2006.
- [22] E. M. Sokhadze, A. El-Baz, J. Baruth, G. Mathai, L. Sears, and M. F. Casanova, "Effects of low frequency repetitive transcranial magnetic stimulation (rTMS) on gamma frequency oscillations and event-related potentials during processing of illusory figures in autism," *J Autism Dev Disord*, vol. 39, pp. 619-34, Apr 2009.
- [23] Y. Bloch, E. V. Harel, S. Aviram, J. Govezensky, G. Ratzoni, and Y. Levkovitz, "Positive effects of repetitive transcranial magnetic stimulation on attention in ADHD Subjects: A

- randomized controlled pilot study," *World Journal of Biological Psychiatry*, vol. 11, pp. 755-758, Aug 2010.
- [24] M. T. Acosta and F. E. Leon-Sarmiento, "Repetitive transcranial magnetic stimulation (rTMS): new tool, new therapy and new hope for ADHD," *Current Medical Research and Opinion*, vol. 19, pp. 125-130, 2003.
- [25] C. S. Konen and P. Haggard, "Multisensory Parietal Cortex contributes to Visual Enhancement of Touch in Humans: A Single-Pulse TMS Study," *Cerebral Cortex*, vol. 24, pp. 501-507, Feb 2014.
- [26] T. Paus, M. A. Castro-Alamancos, and M. Petrides, "Cortico-cortical connectivity of the human mid-dorsolateral frontal cortex and its modulation by repetitive transcranial magnetic stimulation," *European Journal of Neuroscience*, vol. 14, pp. 1405-1411, Oct 2001.
- [27] A. Berardelli, M. Inghilleri, J. C. Rothwell, S. Romeo, A. Curra, F. Gilio, N. Modugno, and M. Manfredi, "Facilitation of muscle evoked responses after repetitive cortical stimulation in man," *Experimental Brain Research*, vol. 122, pp. 79-84, Sep 1998.
- [28] F. Fregni and A. Pascual-Leone, "Transcranial Magnetic Stimulation for the Treatment of Depression in Neurological Disorders", Neuropsychiatric Disorders, pp. 381-390,
- [29] M.C. Eldaief, M.A. Halko, R.L. Buckner, A. Pascual-Leone, Transcranial magnetic stimulation modulates the brain's intrinsic activity in a frequency-dependent manner, Proceedings of the National Academy of Sciences of the United States of America, Vol. 108 (52), pp. 21229-21234, December 2011.
- [30] L. M. Oberman, A Pascual-Leone, A. Rotenberg, "Modulation of corticospinal excitabilty by transcranial magnetic stimulation in children and adolescents with autism spectrum disorder", Frontiers in Human Neuroscience, Vol. 8, August 2014.
- [31] E. M. Wassermann, "Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the international workshop on the safety of repetitive transcranial magnetic stimulation, June 5-7, 1996," *Evoked Potentials-Electroencephalography and Clinical Neurophysiology*, vol. 108, pp. 1-16, Jan 1998.
- [32] S. Rossi, M. Hallett, P. M. Rossini, A. Pascual-Leone, and S. T. C. Grp, "Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research," *Clinical Neurophysiology*, vol. 120, pp. 2008-2039, Dec 2009.

- [33] A.V. Peterchev, T.A Wagner, P.C. Miranda, et al., "Fundamentals of transcranial electric and magnetic stimulation dose: Definition, selection, and reporting practices", Brain Stimulation, Vol. 5 (4) pp. 435-453, October 2012.
- [34] R. Cantello, S. Rossi, C. Varrasi, M. Ulivelli, C. Civardi, S. Bartalini, G. Vatti, M. Cincotta, A. Borgheresi, G. Zaccara, A. Quartarone, D. Crupi, A. Lagana, M. Inghilleri, A. T. Giallonardo, A. Berardelli, L. Pacifici, F. Ferreri, M. Tombini, F. Gilio, P. Quarato, A. Conte, P. Manganotti, L. G. Bongiovanni, F. Monaco, D. Ferrante, and P. M. Rossini, "Slow repetitive TMS for drug-resistant epilepsy: clinical and EEG findings of a placebocontrolled trial," *Epilepsia*, vol. 48, pp. 366-74, Feb 2007.
- [35] F. Fregni, P. T. Otachi, A. Do Valle, P. S. Boggio, G. Thut, S. P. Rigonatti, A. Pascual-Leone, and K. D. Valente, "A randomized clinical trial of repetitive transcranial magnetic stimulation in patients with refractory epilepsy," *Ann Neurol*, vol. 60, pp. 447-55, Oct 2006.
- [36] W. H. Theodore, K. Hunter, R. Chen, F. Vega-Bermudez, B. Boroojerdi, P. Reeves-Tyer, K. Werhahn, K. R. Kelley, and L. Cohen, "Transcranial magnetic stimulation for the treatment of seizures: a controlled study," *Neurology*, vol. 59, pp. 560-2, Aug 27 2002.
- [37] F. Tergau, D. Neumann, F. Rosenow, M. A. Nitsche, W. Paulus, and B. Steinhoff, "Can epilepsies be improved by repetitive transcranial magnetic stimulation?--interim analysis of a controlled study," *Suppl Clin Neurophysiol*, vol. 56, pp. 400-5, 2003.
- [38] J. P. Brasil-Neto, D. P. de Araujo, W. A. Teixeira, V. P. Araujo, and R. Boechat-Barros, "Experimental therapy of epilepsy with transcranial magnetic stimulation Lack of additional benefit with prolonged treatment," *Arquivos De Neuro-Psiquiatria*, vol. 62, pp. 21-25, Mar 2004.
- [39] S. Misawa, S. Kuwabara, K. Shibuya, K. Mamada, and T. Hattori, "Low-frequency transcranial magnetic stimulation for epilepsia partialis continua due to cortical dysplasia," *Journal of the Neurological Sciences*, vol. 234, pp. 37-39, Jul 15 2005.
- [40] D. L. Menkes and M. Gruenthal, "Slow-frequency repetitive transcranial magnetic stimulation in a patient with focal cortical dysplasia," *Epilepsia*, vol. 41, pp. 240-242, Feb 2000.
- [41] S. Rossi, C. Miniussi, P. Pasqualetti, C. Babiloni, P. M. Rossini, and S. F. Cappa, "Agerelated functional changes of prefrontal cortex in long-term memory: A repetitive transcranial magnetic stimulation study," *Journal of Neuroscience*, vol. 24, pp. 7939-7944, Sep 8 2004.
- [42] F. Tergau, U. Naumann, W. Paulus, and B. J. Steinhoff, "Low-frequency repetitive transcranial magnetic stimulation improves intractable epilepsy," *Lancet*, vol. 353, p. 2209, Jun 26 1999.
- [43] M. Kinoshita, A. Ikeda, T. Begum, J. Yamamoto, T. Hitomi, and H. Shibasaki, "Low-frequency repetitive transcranial magnetic stimulation for seizure suppression in patients with extratemporal lobe epilepsy-a pilot study," *Seizure*, vol. 14, pp. 387-92, Sep 2005.
- [44] E. Santiago-Rodriguez, L. Cardenas-Morales, T. Harmony, A. Fernandez-Bouzas, E. Porras-Kattz, and A. Hernandez, "Repetitive transcranial magnetic stimulation decreases

- the number of seizures in patients with focal neocortical epilepsy," *Seizure-European Journal of Epilepsy*, vol. 17, pp. 677-683, Dec 2008.
- [45] H. Quintana, "Transcranial magnetic stimulation in persons younger than the age of 18," *Journal of Ect*, vol. 21, pp. 88-95, Jun 2005.
- [46] K. L. Lin and A. Pascual-Leone, "Transcranial magnetic stimulation and its applications in children," *Chang Gung Med J*, vol. 25, pp. 424-36, Jul 2002.
- [47] R. E. Frye, A. Rotenberg, M. Ousley, and A. Pascual-Leone, "Transcranial Magnetic Stimulation in Child Neurology: Current and Future Directions," *Journal of Child Neurology*, vol. 23, pp. 79-96, Jan 2008.
- [48] K. Muller, V. Homberg, and H. G. Lenard, "Magnetic stimulation of motor cortex and nerve roots in children. Maturation of cortico-motoneuronal projections," *Electroencephalogr Clin Neurophysiol*, vol. 81, pp. 63-70, Feb 1991.
- [49] M. Mohammadi, T. Okanishi, K. Okanari, S. Baba, H. Sumiyoshi, S. Sakuma, A. Ochi, E. Widjaja, C. Y. Go, O. C. Snead, 3rd, and H. Otsubo, "Asymmetrical generalized paroxysmal fast activities in children with intractable localization-related epilepsy," *Brain Dev*, May 5 2014.
- [50] A. Rotenberg, E. H. Bae, P. A. Muller, J. J. Riviello, Jr., B. F. Bourgeois, A. S. Blum, and A. Pascual-Leone, "In-session seizures during low-frequency repetitive transcranial magnetic stimulation in patients with epilepsy," *Epilepsy & Behavior*, vol. 16, pp. 353-5, Oct 2009.
- [51] R. S. Fisher, "Therapeutic devices for epilepsy," *Annals of Neurology*, vol. 71, pp. 157-168, Feb 2012.
- [52] V. K. Kimiskidis, "Transcranial Magnetic Stimulation for Drug-Resistant Epilepsies: Rationale and Clinical Experience," *European Neurology*, vol. 63, pp. 205-210, 2010.
- [53] E. H. Bae, W. H. Theodore, F. Fregni, R. Cantello, A. Pascual-Leone, and A. Rotenberg, "An estimate of placebo effect of repetitive transcranial magnetic stimulation in epilepsy," *Epilepsy & Behavior*, vol. 20, pp. 355-359, Feb 2011.
- [54] F. Cona, M. Zavaglia, M. Massimini, M. Rosanova, and M. Ursino, "A neural mass model of interconnected regions simulates rhythm propagation observed via TMS-EEG," *Neuroimage*, vol. 57, pp. 1045-58, Aug 1 2011.
- [55] F. Farzan, M. A. Halko, A. Pousada-Casal, J. D. Schmahmann, and A. Pascual-Leone, "Modulation and Assessment of the Cerebello-Cortical Connectivity through Transcranial Magnetic Stimulation (TMS) Combined with Electroencephalography (EEG)," *Annals of Neurology*, vol. 72, pp. S82-S83, 2012.
- [56] J. S. Johnson, B. Kundu, A. G. Casali, and B. R. Postle, "Task-dependent changes in cortical excitability and effective connectivity: a combined TMS-EEG study," *Journal of Neurophysiology*, vol. 107, pp. 2383-92, May 2012.
- [57] A. Salah Eddin, J. Wang, W. Wu, S. Sargolzaei, B. Bjornson, R. Jones, W.D. Gaillard, and M. Adjouadi, "The Effects of Pediatric Epilepsy on a Language Connectome", Human

- Brain Mapping, Article first published online: 31 JUL 2014, DOI: 10.1002/hbm.22600, to appear in the December issue Vol. 35 (12), 2014.
- [58] M. Cabrerizo, A. Cabrera, J. Perez, J. De la Rua, N. Rojas, Q. Zhou, A. Pinzon-Ardila, S. Gonzalez-Arias and M. Adjouadi, "Induced Effects of Transcranial Magnetic Stimulation on the Autonomic Nervous System and the Cardiac Rhythm", *Scientific World Journal*, vol. 2014, Article ID 349718, 12 pages, DOI:10.1155/2014/349718, 2014. PMID: 25136660.
- 1) Epilepsy Behav. 2016 Sep;62:136-9. doi: 10.1016/j.yebeh.2016.05.021. Epub 2016 Jul 26. Bursts of high-frequency repetitive transcranial magnetic stimulation (rTMS), together with lorazepam, suppress seizures in a rat kainate status epilepticus model. Gersner R1, Dhamne SC1, Zangen A2, Pascual-Leone A3, Rotenberg A4.
- 2) Epilepsy Res Treat. 2015;2015:678074. doi: 10.1155/2015/678074. Epub 2015 Nov 22. Transcranial Magnetic Stimulation for Status Epilepticus. Zeiler FA1, Matuszczak M2, Teitelbaum J3, Gillman LM4, Kazina CJ1.
- 3) Seizure. 2013 Dec;22(10):893-6. doi: 10.1016/j.seizure.2013.06.014. Epub 2013 Jul 19.Transcranial magnetic stimulation for refractory focal status epilepticus in the intensive care unit.Liu A1, Pang T, Herman S, Pascual-Leone A, Rotenberg A.
- 4) Epilepsy Behav. Author manuscript; available in PMC 2015 Aug 3.Published in final edited form as:Epilepsy Behav. 2009 Jan; 14(1): 253–257.Published online 2008 Oct 30. doi: 10.1016/j.yebeh.2008.09.007PMCID: PMC4523141 NIHMSID: NIHMS92447 PMID: 18832045 Repetitive transcranial magnetic stimulation in treatment of epilepsia partialis continua Alexander Rotenberg, MD, PhD,a,b,\* Erica Hyunji Bae,a Masanori Takeoka,a Jose M. Tormos,b,d Steve C. Schachter,c and Alvaro Pascual-Leone, MD, PhDb,c
- 5) rTMS reduces focal brain hyperperfusion in two patients with EPC. Graff-Guerrero A, Gonzáles-Olvera J, Ruiz-García M, Avila-Ordoñez U, Vaugier V, García-Reyna JC Acta Neurol Scand. 2004 Apr; 109(4):290-6. [PubMed] [Ref list]
- 6) Schrader LMKL, Nuwer MR, Engel J, Stern JM. [Abst. 2.396] Therapeutic efficacy of low frequency repetitive transcranial magnetic stimulation (LF-rTMS) stereotactically directed at a well-defined epileptogenic region (ER). American Epilepsy Society and American Clinical Neurophysiology Society Joint Annual Meeting; 2005; p. 225. [Ref list]
- 7) Misawa S, Kuwabara S, Shibuya K, Mamada K, Hattori T. Low-frequency transcranial magnetic stimulation for epilepsia partialis continua due to cortical dysplasia. J Neurol Sci. 2005;234:37–9.